CLINICAL TRIAL: NCT03143894
Title: Reducing Breast Cancer-related Fatigue and Improving Cognition With Non-Invasive Brain Stimulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual (inability to enroll participants)
Sponsor: Johns Hopkins University (Other)
Collaborators: Under Armour, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00110211; J16135 (Other: Johns Hopkins University)
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Results first posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer; Cognitive Dysfunction; Fatigue
Keywords: Breast Cancer; Cognition; Fatigue; Cancer-related Cognitive Impairment; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction; Fatigue | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized, sham-controlled, double-blind, cross-over
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active tDCS first (Active Comparator): 2 mA of active tDCS applied over a 30-minute study session once per day for 5 consecutive days then sham tDCS after washout.
  Interventions: Device: tDCS; Other: Sham tDCS
- Sham tDCS first (Sham Comparator): Stimulation mimicking the tDCS applied only briefly over a 30-minute study session once per day for 5 consecutive days then active tDCS after washout.
  Interventions: Device: tDCS; Other: Sham tDCS

INTERVENTIONS:
Device: tDCS — Transcranial direct current stimulation (tDCS) is a safe, portable, non-invasive form TDCS is a form of non-invasive electrical brain stimulation using low amplitude direct current to facilitate neuronal transmission beneath scalp electrodes.
  Other Names: Transcranial Direct Current Stimulation; NeuroConn DC Stimulator Plus Model 0021
Other: Sham tDCS — Sham Transcranial direct current stimulation (tDCS)..

SUMMARY:
This study will test the preliminary efficacy of transcranial direct current stimulation (tDCS) to improve fatigue and cognition in women with a history of breast cancer and persistent fatigue.

DETAILED DESCRIPTION:
Fatigue and cognitive dysfunction are commonly reported symptoms associated with impaired quality of life and productivity in breast cancer survivors. Transcranial direct current stimulation (tDCS) has been shown to improve both fatigue and cognition. Here tDCS will be used in a randomized, sham-controlled, double-blind, cross-over trial in women who have finished treatment of breast cancer and who report persistent fatigue.

Participants will complete measures of fatigue and cognition before and after five consecutive days of active or sham tDCS then complete questionnaires by phone one week later. Participants will return about one month later for another five days of participation, followed by another brief study phone call the following week.

ELIGIBILITY:
Inclusion Criteria:

* Women, 18 years of age or older
* Stage I-III breast cancer
* Treatment Status: At least 6 months and no more than 5 years after the conclusion of active breast cancer therapy, including surgery, radiation therapy and (neo)adjuvant chemotherapy, if administered. NOTE: Adjuvant HER2-targeted therapy and endocrine therapy may still be ongoing at the time of study enrollment.
* Fatigue: Moderate fatigue on most days within the past week (i.e., at least 4 out of the last 7 days), rated as ≥ 4 on a 0 (no fatigue) to 10 (worst fatigue) scale.
* Able and willing to complete study tasks as evidenced by at least the following: fluent English speaker; hearing and language comprehension; and, sufficient literacy to complete study forms and questionnaires.
* Patient understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form.

Exclusion Criteria:

* Evidence of recurrent breast cancer at the time of enrollment.
* Depression or anxiety as defined either by ongoing pharmacological treatment for depression or anxiety or a HADS score on initial screening.
* Dementia as assessed by a MMSE score on initial screening.
* Known pregnancy or nursing.
* Any of the following: diagnosis of schizophrenia or bipolar disorder made by a physician, seizure disorder, pacemaker, hearing aids, any metal implanted in the head, or the presence of other known current untreated causes of fatigue such as anemia or untreated hypothyroidism.
* Use of stimulant medications, sleep medications, nicotine patch, and other drugs thought to interfere with tDCS efficacy for seven days prior to and during study participation.
* Use of narcotic pain medication, benzodiazepines, or illicit drugs for seven days prior to and during study participation.
* Consumption of >14 alcoholic drinks per week or positive screening on the CAGE.
* Skin conditions involving open sores on the scalp that would prevent proper application of the electrodes.
* Hairstyles that obstruct placement of the electrodes including cornrows, dreadlocks, braids or other hair accessories that cannot be removed.
* Other medical or other condition(s) that in the opinion of the investigators might compromise the objectives of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-reported gender
Enrollment: 7 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy D Vannorsdall, PhD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins Greenspring Station, Lutherville, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active tDCS First: 2 mA of active tDCS applied over a 30-minute study session once per day for 5 consecutive days. This condition is followed by an active tDCS condition after a washout.
  tDCS: Transcranial direct current stimulation (tDCS) is a safe, portable, non-invasive form TDCS is a form of non-invasive electrical brain stimulation using low amplitude direct current to facilitate neuronal transmission beneath scalp electrodes.
  Sham tDCS: Sham Transcranial direct current stimulation (tDCS).
- Sham tDCS First: Stimulation mimicking the tDCS applied only briefly over a 30-minute study session once per day for 5 consecutive days. This condition is followed by an active tDCS condition after a washout.
  tDCS: Transcranial direct current stimulation (tDCS) is a safe, portable, non-invasive form TDCS is a form of non-invasive electrical brain stimulation using low amplitude direct current to facilitate neuronal transmission beneath scalp electrodes.
  Sham tDCS: Sham Transcranial direct current stimulation (tDCS).
Period: First Intervention (5 Days)
Arm/Group | Active tDCS First | Sham tDCS First
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0
Period: Washout (4 Weeks)
Arm/Group | Active tDCS First | Sham tDCS First
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0
Period: Second Intervention (5 Days)
Arm/Group | Active tDCS First | Sham tDCS First
Started | 3 | 4
Completed | 3 | 3
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS First | Sham tDCS First | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (2.5) | 69 (11.0) | 67.0 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change on Paced Auditory Serial Attention Test (PASAT)
Description: Change in auditory working memory as measured by the PASAT prior to and following the intervention. PASAT scores range from 0 to 120, with higher scores reflecting better working memory. Larger positive change scores reflect greater improvement in performance from baseline whereas greater negative change scores reflect declines in performance from baseline.
Time Frame: Baseline and Day 5
Population: Participants who completed both active and sham conditions, allowing for calculation and comparison of change by condition.
Measure: Mean (Standard Deviation); unit: raw score change on a scale
Groups:
- Active tDCS: 2 mA of active tDCS applied over a 30-minute study session once per day for 5 consecutive days.
  tDCS: Transcranial direct current stimulation (tDCS) is a safe, portable, non-invasive form TDCS is a form of non-invasive electrical brain stimulation using low amplitude direct current to facilitate neuronal transmission beneath scalp electrodes.
  Sham tDCS: Sham Transcranial direct current stimulation (tDCS).
- Sham tDCS: Stimulation mimicking the tDCS applied only briefly over a 30-minute study session once per day for 5 consecutive days.
  tDCS: Transcranial direct current stimulation (tDCS) is a safe, portable, non-invasive form TDCS is a form of non-invasive electrical brain stimulation using low amplitude direct current to facilitate neuronal transmission beneath scalp electrodes.
  Sham tDCS: Sham Transcranial direct current stimulation (tDCS).
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 6 | 6
raw score change on a scale | -1.83 (5.04) | 1.83 (14.52)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; Test type: Superiority; p = 0.47, t-test, 2 sided; Mean Difference (Final Values) = 0.47

2. Secondary Outcome: Change on Functional Assessment of Cancer Therapy Cognitive Scale (FACT-Cog)
Description: Change in subjective cognitive functioning as measured by the FACT-Cog Perceived Cognitive Impairment scale prior to and following the intervention. Raw scores range from 0 to 72, with higher scores reflecting better perceived cognitive functioning. Larger positive change scores reflect greater improvement in subjective cognitive functioning from baseline whereas greater negative change scores reflect declines in subjective cognitive functioning from baseline.
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: raw score change on a scale
Groups:
- Active tDCS (5 Days): 2 mA of active tDCS applied over a 30-minute study session once per day for 5 consecutive days.
  tDCS: Transcranial direct current stimulation (tDCS) is a safe, portable, non-invasive form TDCS is a form of non-invasive electrical brain stimulation using low amplitude direct current to facilitate neuronal transmission beneath scalp electrodes.
  Sham tDCS: Sham Transcranial direct current stimulation (tDCS).
- Sham tDCS (5 Days): Stimulation mimicking the tDCS applied only briefly over a 30-minute study session once per day for 5 consecutive days.
  tDCS: Transcranial direct current stimulation (tDCS) is a safe, portable, non-invasive form TDCS is a form of non-invasive electrical brain stimulation using low amplitude direct current to facilitate neuronal transmission beneath scalp electrodes.
  Sham tDCS: Sham Transcranial direct current stimulation (tDCS).
Arm/Group | Active tDCS (5 Days) | Sham tDCS (5 Days)
Number analyzed (Participants) | 6 | 6
raw score change on a scale | 7.17 (6.55) | 8.67 (12.03)
Statistical Analysis 1: Comparison: Active tDCS (5 Days) vs Sham tDCS (5 Days); Test type: Superiority; p = 0.69, t-test, 2 sided; Mean Difference (Net) = 0.69

3. Secondary Outcome: Change in Multidimensional Fatigue Symptom Inventory- SF (MFSI-SF)
Description: Change in subjective fatigue as measured by the MFSI-SF prior to and following the intervention. Raw scores range from -36 to + 144, with higher scores reflecting greater levels of fatigue. Larger positive change scores reflect greater improvement in fatigue from baseline whereas greater negative change scores reflect declines in fatigue from baseline.
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: raw score change on a scale
Arm/Group | Active tDCS (5 Days) | Sham tDCS (5 Days)
Number analyzed (Participants) | 6 | 6
raw score change on a scale | 8.5 (6.02) | 14.83 (13.69)
Statistical Analysis 1: Comparison: Active tDCS (5 Days) vs Sham tDCS (5 Days); Test type: Superiority; p = 0.36, t-test, 2 sided; Mean Difference (Final Values) = 0.36

ADVERSE EVENTS:
Time Frame: 47 days
Description: Adverse events related to the study intervention were recorded per the descriptions and grading scales found in the revised National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Groups:
- Active tDCS: 2 mA of active tDCS applied over a 30-minute study session once per day for 5 consecutive days.
  tDCS: Transcranial direct current stimulation (tDCS) is a safe, portable, non-invasive form TDCS is a form of non-invasive electrical brain stimulation using low amplitude direct current to facilitate neuronal transmission beneath scalp electrodes.
- Sham tDCS: Stimulation mimicking the tDCS applied only briefly over a 30-minute study session once per day for 5 consecutive days.
  tDCS: Transcranial direct current stimulation (tDCS) is a safe, portable, non-invasive form TDCS is a form of non-invasive electrical brain stimulation using low amplitude direct current to facilitate neuronal transmission beneath scalp electrodes.
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT03143894/Prot_SAP_000.pdf